CLINICAL TRIAL: NCT01407224
Title: Assessing the Cost and Effectiveness of Training and Supervision of Front Line Workers on Early Breastfeeding Practices (Bangladesh)
Brief Title: Assessing Cost and Effectiveness of Training and Supervision of Front Line Workers on Early Breastfeeding Practices
Acronym: iycfch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eminence (Industry)
Collaborators: University of California, Davis (Other)
Responsible Party: Kathyrn Dewey and Shamim Hayder Talukder, UC Davis and Eminence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09-000076-AT10,EMI
Record Dates: First submitted 2011-06-30; First posted 2011-08-02 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Malnutrition
Keywords: Exclusive Breastfeeding; Skin to skin contact; Cord Clumping; Prelactial feeding
MeSH Terms: conditions — Malnutrition; Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Only training (Experimental): Training on Early Breastfeeding Practices to front line health workers
  Interventions: Behavioral: Improve Early Breastfeeding
- Training and supervision (Active Comparator): Training as well as supervision by field supervisor for six months intervention
  Interventions: Behavioral: Improve Early Breastfeeding
- Control (No Intervention): No intervention such as training or supervision
  Interventions: Behavioral: Improve Early Breastfeeding

INTERVENTIONS:
Behavioral: Improve Early Breastfeeding — One arm got only training, another arm training and supervision and third arm without any intervention as control.
  Other Names: IYCFCH

SUMMARY:
The aim of this operational research is to compare the cost-effectiveness of two methods for capacity building of existing TBAs/CVs to improve rates of delayed cord clamping, early skin to skin contact and infant-led initiation of breastfeeding, to reduce prelacteal feeding and increase early exclusive breastfeeding in research areas of rural Bangladesh.

DETAILED DESCRIPTION:
Suboptimal early infant feeding practices are the norm in Bangladesh, and contribute to its poor infant health and nutrition. However, the modern health services are unable to help because approximately 85% of births take place at home. The Government has begun the huge process of training the informal community traditional birth attendants (TBAs) who, along with community volunteers (CVs), deliver the majority of babies, especially in the rural areas. The proposed operations research will take place in one of the poorest rural districts. It will compare the cost effectiveness of practical training of these relatively uneducated community members, with or without supportive supervision in improving early infant feeding practices, using a cluster-randomized study design. The practices to be measured before and after on probability samples include: 1) delayed cord clamping, 2) early skin to skin contact and 3) newborn-led initiation of breastfeeding within one hour of birth, 4) avoidance of the traditional prelacteal feeds, and 5) exclusive breastfeeding, at least for the early months. Costs will be carefully monitored so as to compare the cost per behavior improved per infant.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women of children ages 0 to 5 months and pregnant women with second and third trimester

Exclusion Criteria:

* First trimester women and lactating women of children ages 6 to 23 months.

Ages: 1 Day to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Increased proportions of mothers who follow the recommended infant feeding behaviors | six months intervention
  Practice related to early breastfeeding and cord clumping

SECONDARY OUTCOMES:
Improve practice on breastfeeding, early initiation and cord clumping . | six months intervention
  Evaluation studies are carried out before and after six months of intervention
Improved capacity of TBAs on breastfeeding counseling and knowledge. | Six months
  Increase capacity of TBAs on breastfeeding counseling and knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: DR. Shamim Talukder, M.Phil, Principal Investigator — Eminence
Locations (1):
- Eminence, Dhaka, Bangladesh

REFERENCES:
- [Background] Dewey KG,Talukder S, Greiner T, Farhana D, Shajedul H, Haider R. Assessing cost and effectiveness of training and supervision for front line health workers to improve breastfeeding practice The Lancet 330(13):913-919,2011
- [Derived] Gavine A, Shinwell SC, Buchanan P, Farre A, Wade A, Lynn F, Marshall J, Cumming SE, Dare S, McFadden A. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2022 Oct 25;10(10):CD001141. doi: 10.1002/14651858.CD001141.pub6. PMID 36282618
- See also: RCT of early breastfeeding practices in Bangladesh — http://www.eminence-bd.org